CLINICAL TRIAL: NCT06884267
Title: A Prospective, Multicenter, Single Arm Study to Evaluate the Impact on the Implementation of Standardized Hyperkalemia Management in Chronic Kidney Disease Patients
Brief Title: Hyperkalemia Quality Improvement Program (HK-QIP) Study
Acronym: HK-QIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D9480L00029
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one arm without control group (Other): This is a single-arm interventional study.This study will enroll 1,000 adult Chinese patients with non-dialysis chronic kidney disease (CKD-ND) and HK from around 50 sites in China.
  Interventions: Other: standard hyperkalemia management implementation

INTERVENTIONS:
Other: standard hyperkalemia management implementation — The interventions include HK disease management and quality audits for health care professionals (HCPs) and patients (Figure 1). The main contents of HK disease management in CKD include a standardized clinical pathway based on guideline adoption and medical trainings to educate HCPs and patients.

SUMMARY:
This is a prospective, multi-center, single-arm study to evaluate the impact of implementation of guideline determined medical therapy (GDMT) for quality control improvement in non-dialysis chronic kidney disease (CKD-ND) patients, as well as provide evidence for standard hyperkalemia management with RAASi optimization in China CKD-ND patients.

DETAILED DESCRIPTION:
This is a multi-center, prospective, single-arm interventional study to evaluate the impact on the implementation of standardized hyperkalemia management in CKD patients. Essentially, this is a quality improvement study to determine whether quality improvement intervention can improve medical care process and clinical outcomes.

The intervention of this study is standard hyperkalemia management implementation.

Intervention methods include standard disease management and quality audit.

* Key contents of HK disease management will be standard clinical pathway for management of HK disease based on GDMT (including sK+ > 5.0mmol/L as diagnose criteria; HK long term management; RAASi targeted dose treatment and sK+ test at least once/ 3 months and high-risk patients# once/month). Also track sK+ test frequency and RAASi optimization. Quality audit results as feedback for additional medical education. Medical trainings act as ways to educate HK disease management on both HCPs and patients' level. Education for HCPs include GDMT training*5 times at both study level and individual site level, added at individual site level if quality audit off target (added ≤ 1 time/site quarterly during 0-48 weeks after the first patient enrolled at this site, totally added ≤ 6 times/site). Education for patients include onsite training*6 times during 0-96 weeks and patient self-learning. (# High risk HK patients: CKD with DKD; CKD with HF; CKD with RAASi initiation or up titration.)
* Quality audit includes tracking HCP's perception and action of standardized HK management (quarterly from the first patient enrolled at this site) and patient's adherence to medication and sK+ monitoring (remote visit every 4 weeks [Q4W] and review patient daily checklist every 12 weeks [Q12W]).
* Patient enrolment will begin after the comprehensive GDMT training (both study level and individual site level) for HCPs. Approximately 1,000 adult Chinese patients with renal insufficiency and hyperkalemia will be enrolled from around 50 sites in China. Enrolled patients will be provided with treatment choice and HK management plan determined by HCPs, such as disease education, self management materials, prescription of RAASi use, sK+ test or potassium lowering therapy, etc.
* The follow-up duration will be up to 96 weeks. There will be 6 onsite visits for each patient after baseline visit and data collection, arranged on week 12, week 24, week 36, week 48, week 72 and week 96 after enrolment. Patients who withdraw/discontinue early from the study will have an "early withdrawl" visit.
* There will be remote visit for patients every 4 weeks if no onsite visit after enrolment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, at the time of signing the informed consent.
2. HK (sK+ > 5.0 mmol/L) within 48 hours before enrolment.
3. Patients diagnosed as chronic kidney disease with eGFR>10 ml/min/1.73m2 based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine Equation (2021). See 8.3.4 for detailed equation.
4. Capable of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

1. Patients on dialysis.
2. Pseudohyperkalemia signs and symptoms, such as hemolyzed blood specimen due to excessive fist clenching to make veins prominent, difficult or traumatic venipuncture, or history of severe leukocytosis or thrombocytosis.
3. Patients with acute kidney injury (AKI) or diabetic ketoacidosis (DKA).
4. Patients with cardiac arrhythmias that require immediate treatment
5. Patients scheduled for renal transplant or with a history of renal transplant.
6. Life expectancy < 48 weeks.
7. History of malignancy except for:

   7.1 Malignancy treated with curative intent and with no known active disease within 3 years before the enrolment and of low potential risk for recurrence.

   7.2 Adequately treated non-melanoma skin cancer or lentigo malignancy without evidence of disease.

   7.3 Adequately treated carcinoma in situ without evidence of disease.
8. Be participating in other intervention clinical trials.
9. Judgment by the HCP that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-11-03 (Estimated); Study Completion 2027-11-03 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who achieve RAASi optimizationa with normal sK+ level (3.5 mmol/L ≤ sK+ ≤5.0 mmol/L) after 48 weeks intervention. | Week 48
  To describe the effectiveness of standardized management in patients with CKD and HK for achievement of sK+ control and RAASi optimization

SECONDARY OUTCOMES:
The proportion of patients with normal sK+ level 3.5 mmol/L≤ sK+ ≤ 5.0 mmol/L at each onsite visit. | Week12，Week24，Week36，Week48，Week72，Week96
  To describe the effectiveness of HK standardized management in patients with CKD and HK for achievement of sK+ control
The proportion of patients who achieve RAASi optimization with normal sK+ level (3.5 mmol/L ≤ sK+ ≤ 5.0 mmol/L) after 12 weeks and 24 weeks intervention. | Week12，Week24
  To describe the effectiveness of HK standardized management in patients with CKD and HK for achievement of sK+ control and RAASi optimization during follow up
Percentage change in UACR from baseline to week 48 and week 96 in patients with RAASi use at baseline. | Week48，Week96
  To describe the improvement of urinary albumin after implementation of HK standardized management in patients with CKD and HK

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqiang Ding, Principal Investigator — Fudan University
Locations (39):
- China (39):
  - Research Site, Beijing
  - Research Site, Benxi
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Fuyang
  - Research Site, Fuzhou
  - Research Site, Gejiu
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanning
  - Research Site, Nantong
  - Research Site, Ningbo
  - Research Site, Pingdingshan
  - Research Site, Qiqihar
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Wuhu
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Xining
  - Research Site, Xinxiang
  - Research Site, Yinchuan
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/